CLINICAL TRIAL: NCT02121080
Title: Study of the Safety and Tolerability of REGN2222(SAR438584) in Healthy Adult Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Regeneron Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: R2222-HV-1326
Record Dates: First submitted 2014-04-21; First posted 2014-04-23 (Estimated); Last update posted 2015-03-11 (Estimated); Status verified 2015-03

CONDITIONS: Healthy Volunteers

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (5):
- Cohort 1 (Experimental): Dosing regimen 1
  Interventions: Drug: REGN2222(SAR438584); Drug: placebo
- Cohort 2 (Experimental): Dosing regimen 2
  Interventions: Drug: REGN2222(SAR438584); Drug: placebo
- Cohort 3 (Experimental): Dosing regimen 3
  Interventions: Drug: REGN2222(SAR438584); Drug: placebo
- Cohort 4 (Experimental): Dosing regimen 4
  Interventions: Drug: REGN2222(SAR438584); Drug: placebo
- Cohort 5 (Experimental): Dosing regimen 5
  Interventions: Drug: REGN2222(SAR438584); Drug: placebo

INTERVENTIONS:
Drug: REGN2222(SAR438584)
Drug: placebo

SUMMARY:
This is a phase 1, randomized, double-blind, placebo-controlled study evaluating the safety, tolerability, pharmacokinetic (PK) profile, and immunogenicity of REGN2222 ascending in cohorts of healthy adult volunteers.

ELIGIBILITY:
Inclusion Criteria:

1. A healthy man or woman aged 18 to 60 years
2. Body mass index between 18.0 kg/m2 and 32.0 kg/m2, inclusive
3. Willing and able to comply with clinic visits and study-related procedures
4. Provide signed informed consent

Exclusion Criteria:

1. Serum hemoglobin, creatinine, alkaline phosphatase, CPK, and/or hepatic enzymes (aspartate aminotransferase [AST] and alanine aminotransferase [ALT], total bilirubin [unless the investigator has evidence that increased bilirubin corresponds to a Gilbert's type syndrome with elevated indirect bilirubin]) that is >1.5 the upper limit of normal (ULN), or any laboratory findings showing evidence of organ dysfunction or any clinically significant abnormalities from the normal range, as determined by the investigator at the screening visit
2. Use of any concomitant medications within 30 days or at least 5 half-lives, whichever is longer, of the screening visit, including prescription medications (except contraceptives), nutritional supplements, and over-the-counter medications (except acetaminophen)
3. Hospitalization for any reason within 60 days of the screening visit
4. History of or positive human immunodeficiency virus (HIV) screen result at the screening visit
5. History of or positive blood test result for hepatitis B surface antigen and/or hepatitis C virus antibody at the screening visit
6. History of autoimmune disease
7. History of respiratory disease (e.g, asthma, chronic obstructive pulmonary disease)
8. History of drug or alcohol abuse within 1 year prior to the screening visit
9. Participation in any clinical research study evaluating another investigational drug or therapy within 30 days, or within at least 5 half-lives, of the investigational drug (whichever is longer) prior to the screening visit
10. Pregnant or breastfeeding woman
11. Sexually active men* or women of childbearing potential** who are unwilling to practice adequate contraception during the study, and up to 3 months after the last dose of the study drug (adequate contraceptive measures include stable use of oral contraceptives or other prescription pharmaceutical contraceptives for 2 or more menstrual cycles prior to screening; intrauterine device; bilateral tubal ligation; vasectomy; condom plus contraceptive sponge, foam, or jelly, or diaphragm plus contraceptive sponge, foam, or jelly)

    * Contraception is not required for men with documented vasectomy. **Postmenopausal women must be amenorrheic for at least 12 months in order not to be considered of childbearing potential. Contraception is not required for women with documented hysterectomy or tubal ligation.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 132 (Actual)
Dates: Start 2014-05; Primary Completion 2015-02 (Actual); Study Completion 2015-02 (Actual)

PRIMARY OUTCOMES:
The incidence and severity of treatment-emergent adverse events (TEAEs) in participants treated with REGN2222 or placebo. | from day 1 up to week 20 (EOS)

SECONDARY OUTCOMES:
Serum concentration | from day 1 over time up to week 20
  Serum concentration of REGN2222 over time up to week 20
Presence or absence of antibodies | from day 1 over time up to week 20
  The presence or absence of antibodies against REGN2222 over time up to week 20

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trial Management, Study Director — Regeneron Pharmaceuticals
Locations (3):
- United States (3):
  - Daytona Beach, Florida
  - Evansville, Indiana
  - Dallas, Texas